CLINICAL TRIAL: NCT05033483
Title: Do Iron Supplements Impact the Gut Microbiome of Women of Reproductive Age?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Australian Health and Medical Research Institute (Other)
Collaborators: Flinders University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Iron Mic
Record Dates: First submitted 2021-08-13; First posted 2021-09-02 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2021-11

CONDITIONS: Iron-deficiency; Microbial Colonization; Anemia
Keywords: iron supplements; microbiome; women
MeSH Terms: conditions — Anemia, Iron-Deficiency; Communicable Diseases; Anemia | interventions — ferrous fumarate

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, researcher and participant blinded trial with two parallel groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Supplements were packaged by LifeCare Compounding Pharmacy and labelled by staff not involved in the trial, with 2 colours per treatment group.
  The randomisation schedule was prepared by an independent statistician. The schedule allocates women to one of the four colours in the ratio 1:1:1:1 using randomly permuted blocks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron Supplement (Experimental): 65.7 mg of iron as ferrous fumarate
  Interventions: Dietary Supplement: Ferrous Fumarate
- Placebo (Active Comparator): 0 mg of iron
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ferrous Fumarate — Gelatin capsule containing 200 mg ferrous fumarate and microcrystalline cellulose
  Other Names: Iron Fumarate; ferro-tab
  Arms: Iron Supplement
Dietary Supplement: Placebo — Gelatin capsule containing microcrystalline cellulose
  Other Names: Control
  Arms: Placebo

SUMMARY:
In this randomised controlled trial the investigators will determine whether taking iron supplements compared to placebo for 21 days alters the bacteria (microbiome) in the large intestine of non-pregnant female participants.

DETAILED DESCRIPTION:
BACKGROUND: Many women take iron-containing supplements during pregnancy. Indeed, the World Health Organization recommends that all pregnant women in low-income countries take an iron supplement containing 60 mg/day of elemental iron to reduce iron deficiency and iron-deficiency anaemia. However, oral iron has poor bioavailability, less than 10% absorbed with the remainder passing into the large intestine unbound, potentially providing a competitive advantage to iron-dependent opportunistic pathogens in the large intestine.

In a large randomized control trial in children, iron supplementation was shown to promote the growth of pathogenic species (E. coli, S. aureus, and L. monocytogenes) and inhibited the growth of commensal species (Lactobacillus and Bifidobacterium). These pathogens are associated with enteric infections, while the commensals act on the host's immune system to prevent colonization and invasion by pathogens.

It is NOT known if iron supplementation during pregnancy impacts the maternal and infant microbiome and, by extension, how this affects the neonatal risk of infection and immune dysregulation. Vertical transmission of the maternal microbiome to the newborn is a major determinant of infant health. If maternal iron supplementation affects the infant's health, strategies would be required to mitigate this risk.

The investigators require preliminary data to show how oral iron supplementation alters the intestinal microbiome in women. The Investigators will recruit non-pregnant female participants as there is no risk of vertical transmission to an infant in non-pregnant women. The investigators will conduct the study in Australia because there is not a natural abundance of pathogens that could potentially cause harm to the women. Nevertheless, the investigators would expect a shift in the microbiome from non-iron to iron, requiring bacterial species to return to baseline after women stop taking the iron.

HYPOTHESIS: Daily iron supplementation versus placebo for 21 days will alter the stool microbiome composition compared to placebo in non-pregnant female participants of reproductive age.

METHODS: 80 female participants (18-45 y) will be randomized to receive capsules containing iron (65.7 mg of elemental iron as ferrous fumarate) or placebo to take daily for 21 days. Stool samples will be collected at baseline, 21 days, and 42 days (washout).

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent

Exclusion Criteria:

* Pregnant or breastfeeding.
* Planning on becoming pregnant
* Diagnosed with iron deficiency and/or anaemia in the previous three months
* Taken antibiotics in the past three months
* Taken iron containing supplements in the past three months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Weighted UniFrac dissimilarity score | 21 days
  Measure of microbiota beta-diversity

SECONDARY OUTCOMES:
Bray-Curtis dissimilarity score | 21 days
  Measure of microbiota beta-diversity
Shannon Wiener Diversity | 21 days
  Microbiota alpha-diversity score with adjustment for baseline levels
Faith's phylogenetic diversity | 21 days
  Microbiota alpha-diversity score with adjustment for baseline levels
Taxonomic richness | 21 days
  Microbiota alpha-diversity score with adjustment for baseline levels
Relative abundance of core bacterial taxa | 21 days
  Relative abundance of taxa present in >40% of baseline samples, with adjustment for baseline levels

OTHER OUTCOMES:
Weighted UniFrac dissimilarity score | 42 days (washout)
  Measure of microbiota beta-diversity
Shannon-Wiener diversity | 42 days (washout)
  Microbiota alpha-diversity score with adjustment for baseline levels
Bray-Curtis dissimilarity score | 42 days (washout)
  Measure of microbiota beta-diversity
Faith's phylogenetic diversity | 42 days (washout)
  Microbiota alpha-diversity score with adjustment for baseline levels
Taxonomic richness | 42 days (washout)
  Microbiota alpha-diversity score with adjustment for baseline levels
Relative abundance of core bacterial taxa | 42 days (washout)
  Relative abundance of taxa present in >40% of baseline samples, with adjustment for baseline levels

CONTACTS AND LOCATIONS:
Overall Officials: Steven Taylor, PhD, Principal Investigator — South Australian Health and Medical Research Institute
Locations (1):
- SAHMRI, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
Outlined below
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Following final data analysis and primary publication
Access Criteria: Access to study data may be granted, upon review and approval of the Institutional Review Board, investigators, in accordance with South Australian Health and Medical Research Institute Women and Kids 'Guidelines and Agreement for the use of materials in an ancillary study associated with original clinical trials or cohort studies.

REFERENCES:
- [Derived] Elms L, Hand B, Skubisz M, Best KP, Grzeskowiak LE, Rogers GB, Green TJ, Taylor SL. The Effect of Iron Supplements on the Gut Microbiome of Females of Reproductive Age: A Randomized Controlled Trial. J Nutr. 2024 May;154(5):1582-1587. doi: 10.1016/j.tjnut.2024.03.014. Epub 2024 Mar 21. PMID 38521191